CLINICAL TRIAL: NCT04004299
Title: Time to Diagnosis of HCV Re-infection With the Use of a Self-test: A Feasibility Study
Brief Title: Self-testing for HCV Re-infection in MSM
Acronym: SELFIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Bart Rijnders, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL67745.078.18; MEC-2018-1637 (Other: METC Erasmus MC); IN-NL-987-4653 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2019-06-20; First posted 2019-07-02 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C Recurrent; HIV-1-infection
Keywords: Hepatitis C re-infection

STUDY DESIGN:
Intervention Model Description: Single arm open label multicenter study with diagnostic intervention using capillary blood sampling
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCV self-test intervention (Other): Diagnostic intervention: participant performs capillary blood sampling at home in between outpatient clinic visits (3 months after) and sends the sample to the investigator's laboratory by regular post mail for HCV RNA analysis. This is on top of standard of care ALT measurement at every 6-monthly outpatient clinic visit, followed by HCV RNA testing if ALT is elevated. Follow-up period is 2 years, in which participants will perform and send in 4 self-tests, in combination with filling out 4 questionnaires into sexual risk behavior.
  Interventions: Diagnostic Test: HCV RNA self-test

INTERVENTIONS:
Diagnostic Test: HCV RNA self-test — Self-test set including instruction manual (video available as well), finger prick device, tube and envelope to safely transport biological material. Patient takes capillary blood sample, collects it in the tube and sends the sample to the lab by regular post mail.

SUMMARY:
HIV+MSM (men who have sex with men) that have been cured of a hepatitis C viral infection (HCV) are at risk for HCV re-infection (5-10% per year). One intervention to reduce HCV incidence in this population may be to decrease the time to diagnosis of HCV re-infections in order to decrease the duration that these re-infected patients may transmit their HCV to sex partners. Diagnosis of HCV re-infection is followed by counseling on transmission risk in combination with prompt initiation of HCV therapy, which will prevent new HCV infections on the population level.

In this study the investigators evaluate the effect and feasibility of more frequent and home-based testing for HCV on the time to diagnosis and treatment of HCV re-infections.

DETAILED DESCRIPTION:
Elimination of HCV was recently formulated as a WHO target and was set for the year 2030. Globally, approximately 6.2% of HIV-infected patients are co-infected with HCV. Of the patients living with HIV, people who inject drugs (PWID) and men who have sex with men (MSM) are at particularly high risk of HCV co-infection. Until recently, the prevalence of chronic hepatitis C virus infection (HCV) in Dutch HIV+MSM was very high at 4,8% (compared with 0.2% in the Dutch population in general). After unrestricted availability of direct-acting antivirals since the end of 2015, the prevalence of chronic HCV in HIV+MSM decreased rapidly. A subsequent decrease in the incidence of HCV of 51% was observed in 2016, but no further decline was seen in 2017. Additionally, the incidence of HCV re-infections in HIV+MSM that were cured of a previous HCV infection continues to be high (5-10% per year).

The continuously high re-infection risk and the lack of a further decline in the HCV incidence after 2016 illustrates that universal DAA therapy for all patients diagnosed with a chronic HCV infection on its own will not result in HCV elimination. Other interventions are needed to reach the WHO goal of HCV elimination by 2030. One of these additional interventions may be decreasing the time to diagnosis of HCV re-infections in order to decrease the duration that these re-infected patients may transmit their HCV to sex partners.

Objective:

To assess the effectivity of HCV RNA self-testing in reducing the time to diagnosis of HCV re-infection in MSM previously cured of an HCV infection, compared to the current diagnostic standard of care.

To evaluate whether the uptake of self-testing is sufficient and warrants the use of HCV RNA self-testing in clinical practice.

Study design:

Prospective controlled intervention trial. MSM cured of an HCV infection who are at continued risk for an HCV re-infection (based on the results of a short questionnaire, APPENDIX B) are offered HCV RNA self-testing and asked to use the test every 6 months for 2 consecutive years.

Study population:

225 to 250 adult MSM cured of HCV from 10-15 HIV and PREP clinics in the Netherlands and Belgium.

Intervention:

Eligible patients are instructed on the use of a capillary blood self-collection kit. They receive 2 kits per year for 2 consecutive years to allow them to send plasma to the virology lab of the Erasmus MC every 6 months by regular post mail.

Primary endpoints:

Comparison of the time to HCV re-infection diagnosis in patients using the HCV RNA self-test (intervention) with the time to HCV re-infection diagnosis with the standard diagnostic approach (control) in the modified intention to treat population.

Secondary endpoints:

1. Comparison of the time to HCV re-infection diagnosis in patients using the HCV RNA self-test (intervention) with the time to HCV re-infection diagnosis with the standard diagnostic approach (control) in the subpopulation that has sent in all planned self-tests during their entire follow-up (per protocol analysis).
2. Of the HIV+MSM that were offered to participate in the study, the percentage that accepted to participate and eventually self-collected and sent in at least one plasma sample in each 12-month period of study participation.
3. Overall incidence of HCV re-infection in the entire study population regardless of the type HCV diagnostic test that was used.
4. Number of screen failures as a result of a positive HCV-RNA test at the screening visit.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The burden associated with participation in the study consists of taking a finger prick blood sample for the self-test 4 times in 2 years and sending the sample to the laboratory by regular post mail. No costs will have to be made for mailing the sample. Capillary finger-prick blood sampling is used as a standard diagnostic test for many diseases (e.g. glucose monitoring in diabetes) and is associated with a negligible risk. The study may potentially be beneficial for those participants in which an HCV re-infection is diagnosed as they will be referred for counseling and HCV therapy which has the potential to prevent transmission to sex partners.

ELIGIBILITY:
Inclusion Criteria:

* Cured of HCV defined as an SVR (=documented negative HCV RNA test) at least 12 weeks after the end of DAA therapy and no new documented positive HCV RNA test after the date of the SVR

OR

Spontaneous clearance of HCV infection defined as two consecutive negative HCV RNA tests at least 3 months apart after a positive HCV RNA test.

* In care for an HIV infection in an HIV clinic in a study center or HIV negative and receiving PrEP at a PrEP clinic
* Able and willing to perform the self-test at home after viewing the instruction video
* Willing to fill out a questionnaire on risk behavior at the time of HCV self-testing
* At risk of HCV re-infection according to a short questionnaire, in other words, patients should have one of the following risk factors:

  * Receptive unprotected (condomless) anal intercourse in the last 6 months
  * Fisting or being fisted without gloves in the last 6 months
  * Sharing toys in the last 6 months
  * Syphilis or LGV in the last 12 months,
  * Slamming (injecting drug use) in the last 12 months
  * Sharing sniffing straws or other objects to sniff drugs in the last 12 months

Exclusion Criteria:

* Age < 18
* Patients that are tested by HCV RNA as a standard of care test (e.g. in the context of PREP use) > 1x/year
* Patients that are expected to be tested by ALT at their HIV or PREP clinic <1x/year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in time to HCV re-infection diagnosis with the intervention in MITT population | Last negative HCV test to first positive HCV test (from start study to first positive HCV test in up to 2 years)
  Comparison of the time to HCV re-infection diagnosis in patients using the HCV RNA self-test (intervention) with the time to HCV re-infection diagnosis with the standard diagnostic approach (virtual control) in the modified intention to treat (MITT) population.

SECONDARY OUTCOMES:
Change in time to HCV re-infection diagnosis with the intervention in PP | Last negative HCV test to first positive HCV test (from start study to first positive HCV test in up to 2 years)
  Comparison of the time to HCV re-infection diagnosis in patients using the HCV RNA self-test (intervention) with the time to HCV re-infection diagnosis with the standard diagnostic approach (virtual control) in the subpopulation that sent in all planned self-tests during their entire follow-up (Per Protocol analysis).
Acceptability of intervention in target population: percentage that accepted to participate and eventually self-collected and sent in at least one plasma sample | Through study process, from start screening to study completion, at least 3 years
  Of the HIV+MSM that were offered to participate in the study, the percentage that accepted to participate and eventually self-collected and sent in at least one plasma sample in each 12-month period of study participation.
HCV re-infection incidence in study population | During follow-up period of 2 years
  Overall incidence of HCV re-infection in the entire study population regardless of the type of HCV diagnostic test that was used.
HCV infections found at screening | At screening visit (T=0)
  Number of newly diagnosed HCV infections at the time of the screening visit as a result of a positive HCV-RNA test at the screening visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Rijnders, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (7):
- Netherlands (7):
  - Ziekenhuis Rijnstate, Arnhem, Gelderland
  - Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Spaarne Gasthuis, Haarlem, South Holland
  - Erasmus Medical Center (EMC), Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Utrecht Medical University Center (UMCU), Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boerekamps A, van den Berk GE, Lauw FN, Leyten EM, van Kasteren ME, van Eeden A, Posthouwer D, Claassen MA, Dofferhoff AS, Verhagen DWM, Bierman WF, Lettinga KD, Kroon FP, Delsing CE, Groeneveld PH, Soetekouw R, Peters EJ, Hullegie SJ, Popping S, van de Vijver DAMC, Boucher CA, Arends JE, Rijnders BJ. Declining Hepatitis C Virus (HCV) Incidence in Dutch Human Immunodeficiency Virus-Positive Men Who Have Sex With Men After Unrestricted Access to HCV Therapy. Clin Infect Dis. 2018 Apr 17;66(9):1360-1365. doi: 10.1093/cid/cix1007. PMID 29186320
- [Background] Ingiliz P, Martin TC, Rodger A, Stellbrink HJ, Mauss S, Boesecke C, Mandorfer M, Bottero J, Baumgarten A, Bhagani S, Lacombe K, Nelson M, Rockstroh JK; NEAT study group. HCV reinfection incidence and spontaneous clearance rates in HIV-positive men who have sex with men in Western Europe. J Hepatol. 2017 Feb;66(2):282-287. doi: 10.1016/j.jhep.2016.09.004. Epub 2016 Sep 17. PMID 27650285
- [Background] Vanhommerig JW, Lambers FA, Schinkel J, Geskus RB, Arends JE, van de Laar TJ, Lauw FN, Brinkman K, Gras L, Rijnders BJ, van der Meer JT, Prins M; MOSAIC (MSM Observational Study of Acute Infection With Hepatitis C) Study Group; van der Meer JT, Molenkamp R, Mutschelknauss M, Nobel HE, Reesink HW, Schinkel J, van der Valk M, van den Berk GE, Brinkman K, Kwa D, van der Meche N, Toonen A, Vos D, van Broekhuizen M, Lauw FN, Mulder JW, Arends JE, van Kessel A, de Kroon I, Boonstra A, van der Ende ME, Hullegie S, Rijnders BJ, van de Laar TJ, Gras L, Smit C, Lambers FA, Prins M, Vanhommerig JW, van der Veldt W. Risk Factors for Sexual Transmission of Hepatitis C Virus Among Human Immunodeficiency Virus-Infected Men Who Have Sex With Men: A Case-Control Study. Open Forum Infect Dis. 2015 Aug 6;2(3):ofv115. doi: 10.1093/ofid/ofv115. eCollection 2015 Sep. PMID 26634219

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT04004299/Prot_SAP_000.pdf